CLINICAL TRIAL: NCT06798506
Title: A Real-world, Multicenter, Prospective Study to Evaluate the Patient-reported Outcome in Chinese Patients Who Received Sacituzumab Govitecan or Chemotherapy of the Physician's Choice for Metastatic Triple-negative Breast Cancer
Brief Title: Real-world Patient-reported Outcome of Sacituzumab Govitecan in Chinese Metastatic Triple-negative Breast Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Biyun Wang, MD, Professor, Fudan University
Other Study IDs: YOUNGBC-32
Record Dates: First submitted 2024-12-18; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-12

CONDITIONS: TNBC - Triple-Negative Breast Cancer
Keywords: Sacituzumab Govitecan; chemotherapy; metastatic breast cancer; TNBC
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Sacituzumab Govitecan cohort
- Chemotherapy of the physician's choice cohort

SUMMARY:
The aim of this trial is to explore the real-world patient-reported health-related quality of life (HRQOL), functioning, symptoms and symptom tolerability of sacituzumab govitecan or chemotherapy of the physician's choice for Chinese mTNBC patients. Evaluation of HRQOL and functioning using the EORTC QLQ-C30 and QLQ-BR45 questionnaires, including change from baseline and time to deterioration in each scale or item. Treatment-related symptoms and tolerability were assessed using the Patient-Reported Outcomes of the PRO-CTCAE and PGI-TT questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged over 18 years old.
2. Patients have been diagnosed with metastatic triple-negative breast cancer (mTNBC). ER, PgR, and HER2 status were determined locally by immunohistochemistry (IHC) of patients' primary or metastatic tumor sections. ER-negative and PgR-negative status was defined as≤1% staining in the nuclei by IHC. HER2-negative status was defined by IHC staining 0 to 1+ or fluorescence in situ hybridization ratio <2.0 if IHC 2+ or IHC not performed.
3. The metastatic disease was confirmed by clinical, imaging, histological, or cytological measures, including unresectable locally advanced breast cancer, de novo stage IV breast cancer, and recurrent metastatic breast cancer.
4. Patients who have received at least 1 prior regimen in the metastatic setting.
5. Plan to receive or has received sacituzumab govitecan monotherapy or chemotherapy of the physician's choice.
6. Available medical history.
7. All patients can provide an informed consent before enrolment and data collection.

Exclusion Criteria:

1. If participating in any controlled clinical trial, the subject cannot take part in this study.
2. HER2 overexpression or gene amplification, ie, immunohistochemistry (IHC) 3+ or fluorescence in situ hybridisation (FISH)+, where appropriate.
3. Pregnancy and lactation.
4. Severe hepatic impairment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients have been diagnosed with metastatic triple-negative breast cancer (mTNBC). ER, PgR, and HER2 status were determined locally by immunohistochemistry (IHC) of patients' primary or metastatic tumor sections.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-05-15 (Estimated)

PRIMARY OUTCOMES:
Patient-reported HRQOL | 6 weeks
  Patient-reported health-related quality of life (HRQOL) evaluated by EORTC QLQ-C30 questionnaires

SECONDARY OUTCOMES:
Patient-reported functioning | 6 weeks
  Patient-reported functioning evaluated by QLQ-BR45 questionnaires.
Patient-reported symptoms | 6 weeks
  Treatment-related symptoms were assessed using the Patient-Reported Outcomes of the PRO-CTCAE.
Patient-reported tolerability | 6 weeks
  Treatment-related tolerability were assessed using the Patient-Reported Outcomes of the PGI-TT questionnaires.
PFS | 6 weeks
  Progression free survival
ORR | 6 weeks
  Overall Response Rate
CBR | 6 weeks
  Clinical benefit Rates
OS | 6 weeks
  Overall Survival
Safety | 6 weeks
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China